CLINICAL TRIAL: NCT04491838
Title: A Randomized, Open-Label, Parallel Group Study of the Pharmacokinetics, Safety, and Tolerability of a Single Subcutaneous Dose of Pozelimab Produced From Two Different Manufacturing Processes in Healthy Subjects
Brief Title: Study of a Single Subcutaneous Dose of Pozelimab Produced From Two Different Manufacturing Processes in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3918-HV-2014; 2020-002365-33 (EudraCT Number)
Record Dates: First submitted 2020-07-13; First posted 2020-07-29 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Process A (Experimental): Randomized 1:1
  Interventions: Drug: Pozelimab
- Process B (Experimental): Randomized 1:1
  Interventions: Drug: Pozelimab

INTERVENTIONS:
Drug: Pozelimab — Single subcutaneous (SC) injection
  Other Names: REGN3918

SUMMARY:
The primary objective of the study is to compare the pharmacokinetic(PK) profile of pozelimab produced by the original manufacturing process (Process A) compared to a second manufacturing process (Process B)

The secondary objectives of the study are:

* Assess the safety and tolerability of a single SC dose of pozelimab produced by the 2 manufacturing processes
* Assess the immunogenicity of pozelimab produced by the 2 manufacturing processes

ELIGIBILITY:
Key Inclusion Criteria:

* Has a body weight of 55 kg to 100 kg and a body mass index between 18 kg/m2 and 30 kg/m2 inclusive at the screening visit
* Judged to be in good health based on medical history, physical examination, vital signs measurements, and ECG performed at screening and/or prior to administration of initial dose of study drug
* Is in good health based on laboratory safety testing obtained at the screening visit. NOTE: Subject with a history of Gilbert's disease can be enrolled in the study
* Willing to undergo vaccination against N meningitidis unless subjects have documentation of completed series of vaccinations within the past 2 years of the screening visit
* Must have two negative COVID-19 tests within 7 days prior to study drug administration as defined in the protocol

Key Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease, as assessed by the investigator
* Hospitalization (>24 h) for any reason within 90 days of the screening visit
* Has a confirmed positive drug test result at the screening visit and/or prior to enrollment; and/or a history of recreational drug use (eg, marijuana) and/or drug or alcohol abuse within a year prior to the screening visit
* Is positive for HIV, hepatitis B, or hepatitis C antibody as defined in the protocol
* Known or suspected COVID-19 disease
* History of tuberculosis, systemic fungal diseases, or meningococcal infection
* Known allergy or intolerance to penicillin class antibiotics or macrolides; any contraindication to azrithromycin per local prescribing information

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Assess the time of the last positive concentration (AUClast) pharmacokinetic (PK) profile of pozelimab in Process A | Up to 16 weeks
Assess the time of the last positive concentration (AUClast) PK profile of pozelimab in Process B | Up to 16 weeks
Assess peak concentration (Cmax) PK profile of pozelimabin in Process A | Up to 16 weeks
Assess peak concentration (Cmax) PK profile of pozelimab in Process B | Up to 16 weeks

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to 16 weeks
Incidence of anti-drug antibodies (ADA) to pozelimab over time | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Study Site, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/